CLINICAL TRIAL: NCT05614089
Title: Human Versus Analogue Insulin for Youth With Type 1 Diabetes in Low-Resource Settings: A Randomized Controlled Trial
Brief Title: Human Versus Analogue Insulin for Youth With Type 1 Diabetes in Low-Resource Settings
Acronym: HumAn-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jing Luo (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor-Investigator, Jing Luo, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY21110122
Record Dates: First submitted 2022-10-28; First posted 2022-11-14 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1; Type 1 Diabetes
Keywords: Type 1 Diabetes; Insulin Glargine; Human Insulin; Insulin Analogue; Bangladesh; Tanzania
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin Glargine; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Glargine (Experimental): Insulin glargine (long-acting insulin analogue)
  Interventions: Drug: Insulin Glargine
- NPH or premixed 70/30 (human insulin) (Active Comparator): NPH or premixed 70/30 (human insulin)
  Interventions: Drug: NPH or premixed 70/30 (human insulin)

INTERVENTIONS:
Drug: Insulin Glargine — Formulation: Available as a clear liquid in a glass cartridge (1 cartridge =3ml=300 units).
  Route: Reusable pen
  Amount of each dose: varies depending on baseline basal insulin needs
  Dose escalation scheme: Participants randomly assigned to glargine will start with a dose that is generally equal to 80% of their total basal human insulin dose prior to the switch (per ISPAD guidelines and the switching guide developed by Life for a Child with the guidance of Dr. Ragnar Hanas and two other ISPAD members familiar with less-resourced settings).
  Frequency of dose: once per day (usually administered before bedtime)
  Duration of therapy: 12 months
  Arms: Glargine
Drug: NPH or premixed 70/30 (human insulin) — Formulation: Available as a liquid in a glass cartridge (3ml=300IU) or as liquid in a prefilled, disposable pen (3ml=300IU).
  Route: Bangladesh = reusable pens; Tanzania = disposable pens
  Amount of each dose: varies depending on baseline basal insulin needs (per usual care or treating clinician)
  Frequency of dose: once or twice per day (per usual care or treating clinician)
  Duration of therapy: 12 months
  Arms: NPH or premixed 70/30 (human insulin)

SUMMARY:
The primary objective of this trial is to determine whether insulin glargine reduces the risk of serious hypoglycemia or improves Time in Range at 6 months when compared against standard of care human insulin (e.g. NPH or premixed 70/30) among youth living with type 1 diabetes (T1D) in low resource settings.

DETAILED DESCRIPTION:
Long-acting insulin analogues have become a de-facto standard of care for patients with T1D living in high-income countries. Unfortunately, insulin analogues remain unavailable or unaffordable for much of the global population. In both 2017 and 2019, applications to add long-acting insulin analogues to the WHO's Model List of Essential Medicines (EML) were rejected due to insufficient evidence of superiority and an unfavorable cost-effectiveness profile when compared against older, less expensive, human insulins (e.g., NPH insulin and premixed 70/30 insulin). In 2021, long-acting insulin analogues were added to the EML but the decision remains controversial since the WHO concluded that "magnitude of clinical benefit of long-acting insulin analogues over human insulin for most clinical outcomes was small." Moreover, studies that compare long-acting insulin analogues versus human insulins conducted in high-income settings may not generalize to children and young adults living with T1D in very low-resource settings.

To address this unmet need, Pitt has partnered with Brigham and Women's Hospital, The London School of Hygiene and Tropical Medicine, the Clinton Health Access Initiative and Life For a Child to conduct a randomized controlled trial comparing insulin glargine, a long-acting analogue insulin, against intermediate human insulin among 400 children and young adults living with T1D in a lower resource setting.

Note: In preparation for results submission, we made minor changes to the outcomes sections to reflect what is listed in the protocol.

For Primary Outcomes #1 and #2, and Secondary Outcomes #3,#4, #5, #7, #8: we added 12 months measurements (in addition to the 6 months measurement). We updated Secondary Outcome #9 to specify the PedsQL Diabetes Symptoms Score. We added Secondary Outcome #10 to include the PedsQL Diabetes Management Score. We added Secondary Outcome #11 for ITSQ scores.

ELIGIBILITY:
Inclusion Criteria:

1. Children and young adults (age 7-25)
2. Have a clinical diagnosis of type 1 diabetes (T1D)

Exclusion Criteria:

1. Prior use of any insulin analogue
2. Patients (or parents for children <18 years old) who refuse to or cannot provide informed consent
3. Who are currently pregnant or plan to become pregnant over the next year
4. Who have previously used a continuous glucose monitor (CGM) for glucose monitoring
5. Who were first diagnosed with T1D less than 12 months ago
6. Who is diagnosed with severe malnutrition

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2025-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Luo, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (3):
- BIRDEM Hospital, Dhaka, Bangladesh
- Tanzania (2):
  - Bugando Medical Center, Mwanza
  - Sekou-Toure Hospital, Mwanza

IPD SHARING:
Plan to Share IPD: Yes
De-identified, summary level data will be shared with other researchers, upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 3 years after the completion of the primary endpoint (Start 16 September 2024; End 16 September 2027)
Access Criteria: Researchers who provide a methodologically sound proposal, upon request

REFERENCES:
- [Derived] Foulds A, Josey C, Kehlenbrink S, Rollman BL, Chang CH, Lalama C, Ansbro E, Prust ML, Zabeen B, Ramaiya K, Ogle G, Chae SR, Luo J. Human versus Analogue Insulin for Youth with Type 1 Diabetes in Low-Resource Settings (HumAn-1): protocol for a randomised controlled trial. BMJ Open. 2025 Jan 30;15(1):e092432. doi: 10.1136/bmjopen-2024-092432. PMID 39890140

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants consented and had baseline demographics collected in-person and/or baseline/run-in CGM placed, but withdrew from study before randomization to arm due to the following reasons: No longer interested in participating, Became ineligible
Groups:
- Glargine: Insulin glargine (long-acting insulin analogue)
  Insulin Glargine: Formulation: Available as a clear liquid in a glass cartridge (1 cartridge =3ml=300 units).
  Route: Reusable pen
  Amount of each dose: varies depending on baseline basal insulin needs
  Dose escalation scheme: Participants randomly assigned to glargine will start with a dose that is generally equal to 80% of their total basal human insulin dose prior to the switch (per ISPAD guidelines and the switching guide developed by Life for a Child with the guidance of Dr. Ragnar Hanas and two other ISPAD members familiar with less-resourced settings).
  Frequency of dose: once per day (usually administered before bedtime)
  Duration of therapy: 12 months
- NPH or Premixed 70/30 (Human Insulin): NPH or premixed 70/30 (human insulin)
  NPH or premixed 70/30 (human insulin): Formulation: Available as a liquid in a glass vial or glass cartridge (10ml=1000IU).
  Route: Bangladesh = syringes or reusable pens; Tanzania = disposable pens
  Subcutaneous injection using insulin syringe and needle
  Amount of each dose: varies depending on baseline basal insulin needs (per usual care or treating clinician)
  Frequency of dose: once or twice per day (per usual care or treating clinician)
  Duration of therapy: 12 months
Period: Overall Study
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Started | 199 | 201
Clinic Visit 2 (6-months) (When a first primary endpoint CGM is placed and HbA1c collected) | 196 | 199
Home Visit 2 (6.5-months) (When clinic visit 2 (6-month) CGM is removed/data collected and second primary endpoint CGM is placed) | 196 | 199
Home Visit 3 (7-months) (When home visit 2 (6.5-month) CGM is removed/data collected) | 196 | 199
Completed | 188 | 197
Not Completed | 11 | 4
Not completed — Pregnancy | 5 | 2
Not completed — Lost to Follow-up | 5 | 1
Not completed — Death | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin) | Total
Number analyzed (Participants) | 199 | 201 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.1 (5.2) | 16.6 (5.0) | 16.8 (5.1)
Age, Customized [Count of Participants; unit: Participants]
  Age, categorical: 7 -<10 years | 26 | 24 | 50
  Age, categorical: 10 -<18 years | 84 | 88 | 172
  Age, categorical: 18 - <26 years | 89 | 89 | 178
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 115 | 222
  Male | 92 | 86 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity/Tribe: Bengali | 124 | 126 | 250
  Ethnicity/Tribe: Sukuma | 41 | 47 | 88
  Ethnicity/Tribe: Kurya | 4 | 4 | 8
  Ethnicity/Tribe: Haya | 2 | 4 | 6
  Ethnicity/Tribe: Other | 28 | 20 | 48
Region of Enrollment [Number; unit: participants]
  Bangladesh | 124 | 126 | 250
  Tanzania | 75 | 75 | 150
BMI [Mean (Standard Deviation); unit: (kg/m^2)] | 20.3 (4.0) | 19.8 (3.7) | 20.0 (3.9)
Education of Participant [Count of Participants; unit: Participants]
  University | 14 | 11 | 25
  College/Diploma | 44 | 54 | 98
  Secondary School/Education | 76 | 67 | 143
  Primary School/Education | 64 | 66 | 130
  No Education | 1 | 3 | 4
Education of Parent [Count of Participants; unit: Participants]
  University | 23 | 26 | 49
  College/Diploma | 26 | 36 | 62
  Secondary School/Education | 93 | 77 | 170
  Primary School/Education | 47 | 46 | 93
  No Education | 10 | 14 | 24
  Don't know | 0 | 2 | 2
# of Adults Living with [Mean (Standard Deviation); unit: number of people] | 3.1 (1.8) | 2.8 (1.3) | 2.9 (1.6)
Socioeconomic Status [Count of Participants; unit: Participants]
  Poor | 97 | 96 | 193
  Lower middle | 33 | 29 | 62
  Middle | 60 | 63 | 123
  Upper middle | 6 | 12 | 18
  Rice farmer | 1 | 0 | 1
  Well off/Rich | 2 | 1 | 3
Duration of Type 1 Diabetes [Mean (Standard Deviation); unit: years] | 5.9 (4.2) | 5.9 (3.8) | 5.9 (4.0)
Type of Insulin Regimen [Count of Participants; unit: Participants]
  NPH + Regular with meals | 196 | 196 | 392
  Premixed 70/30 alone | 3 | 3 | 6
  Premixed 70/30 + Regular with meals | 0 | 2 | 2
Total Number of Units of Insulin per Day/Weight [Mean (Standard Deviation); unit: insulin units/kg per day] | 1.0 (0.4) | 1.1 (0.4) | 1.0 (0.4)
HbA1c [Mean (Standard Deviation); unit: percent] | 9.7 (2.8) | 9.9 (2.8) | 9.8 (2.8)
c-peptide [Mean (Standard Deviation); unit: ng/mL] — Population: Twenty-three (23) and 26 participants, respectively, had results below the limit, and lab not done in 3 participants in the glargine group.
  ng/mL
    number analyzed (Participants) | 173 | 175 | 348
    (all) | 0.25 (0.31) | 0.25 (0.34) | 0.25 (0.32)
History of DKA (diabetic ketoacidosis) [Count of Participants; unit: Participants]
  Yes | 53 | 61 | 114
  No | 146 | 139 | 285
  Don't know | 0 | 1 | 1
Number of Severe Hypoglycemic Events [Mean (Standard Deviation); unit: number of events] — Severe hypoglycemic events (requiring assistance of another person to correct) in past 12 months reported by participant Population: One participant in each arm did not know the number of severe hypoglycemic events they had in past 12 months
  number of events
    number analyzed (Participants) | 198 | 200 | 398
    (all) | 0.9 (1.9) | 0.8 (1.7) | 0.9 (1.8)
Number of Symptomatic Hypoglycemic Events [Mean (Standard Deviation); unit: number of events] — Symptomatic hypoglycemic events (e.g. dizziness, confusion) in past 30 days reported by participant Population: Eleven (11) and 7 participants, respectively, did not know the number of symptomatic hypoglycemic events they had in past 30 days
  number of events
    number analyzed (Participants) | 188 | 194 | 382
    (all) | 1.9 (2.4) | 2.0 (2.6) | 1.9 (2.5)
Number of Asymptomatic Hypoglycemic Events [Mean (Standard Deviation); unit: number of events] — Asymptomatic hypoglycemic events (i.e. blood glucose < 3.9 mmol/L (70mg/dl) without clinical symptoms) in past 30 days reported by participant Population: Twenty-one (21) and 7 participants, respectively, did not know the number of asymptomatic hypoglycemic events they had in past 30 days
  number of events
    number analyzed (Participants) | 178 | 194 | 372
    (all) | 1.0 (2.4) | 1.1 (1.9) | 1.0 (2.1)
Retinopathy [Count of Participants; unit: Participants] — Diabetes comorbidities from medical record
  Participants | 8 | 6 | 14
Nephropathy [Count of Participants; unit: Participants] — Diabetes comorbidities from medical record
  Participants | 2 | 3 | 5
Diabetic Foot Disease [Count of Participants; unit: Participants] — Diabetes comorbidities from medical record
  Participants | 2 | 0 | 2
Amputation [Count of Participants; unit: Participants] — Diabetes comorbidities from medical record
  Participants | 0 | 0 | 0
Neuropathy [Count of Participants; unit: Participants] — Diabetes comorbidities from medical record
  Participants | 3 | 1 | 4
Percent Time in Serious Hypoglycemia [Mean (Standard Deviation); unit: percentage of time] — Percent time in serious hypoglycemia (<54 mg/dl) averaged across all daily measures from CGM placed at baseline and worn during run-in phase
  percentage of time | 3.7 (5.0) | 3.7 (5.6) | 3.7 (5.3)
Percent Time in Range [Mean (Standard Deviation); unit: percentage of time] — Percent time in glycemic range (70-180 mg/dL, inclusive) averaged across all daily measures from CGM placed at baseline and worn during run-in phase
  percentage of time | 38.9 (20.9) | 35.0 (19.3) | 36.9 (20.1)
Percent Time in Hypoglycemia [Mean (Standard Deviation); unit: percentage of time] — Percent time below glycemic range (<70 mg/dl) averaged across all daily measures from CGM placed at baseline and worn during run-in phase
  percentage of time | 10.9 (10.2) | 10.7 (11.2) | 10.8 (10.7)
Percent Time Above Range [Mean (Standard Deviation); unit: percentage of time] — Percent time above glycemic range (>180 mg/dl) averaged across all daily measures from CGM placed at baseline and worn during run-in phase
  percentage of time | 50.2 (26.7) | 54.3 (26.6) | 52.3 (26.7)
Nocturnal Hypoglycemic Events [Mean (Standard Deviation); unit: number of events] — Events are defined as ≥15 minutes in duration <70 mg/dL between midnight and 6:00 am; specifically, at least 2 sensor values <70 mg/dL (from CGM placed at baseline and worn during run-in phase) that are ≥15 minutes apart plus no intervening values ≥70 mg/dL Population: For 3 participants in each arm, the CGM only had 1 active day and did not have any data during the nocturnal hours
  number of events
    number analyzed (Participants) | 196 | 198 | 394
    (all) | 3.6 (3.4) | 3.4 (3.2) | 3.5 (3.3)
Pediatric Quality of Life Inventory 3.2 Diabetes Module (PedsQL 3.2 DM) Diabetes Symptoms Score [Mean (Standard Deviation); unit: score on a scale] — PedsQL 3.2 DM Diabetes Symptoms scale is composed of 15 items. All items use the same 5-point Likert response scale, with responses ranging from "never" (0) to "almost always" (4). Items are reverse scored and transformed on a scale ranging from 0 to 100. The score is the sum of all the items over the number of items answered. Higher scores indicate fewer diabetes symptoms and therefore improved D-HRQoL.
  score on a scale | 68.1 (14.7) | 69.3 (14.0) | 68.7 (14.4)
Pediatric Quality of Life Inventory 3.2 Diabetes Module (PedsQL 3.2 DM) Diabetes Management Score [Mean (Standard Deviation); unit: score on a scale] — PedsQL 3.2 DM Diabetes Management scale is composed of 18 items. All items use the same 5-point Likert response scale, with responses ranging from "never" (0) to "almost always" (4). Items are reverse scored and transformed on a scale ranging from 0 to 100. Higher scores indicate fewer diabetes management problems and therefore improved D-HRQoL.
  score on a scale | 80.0 (14.3) | 81.5 (13.8) | 80.7 (14.0)
ITSQ Total [Mean (Standard Deviation); unit: score on a scale] — The ITSQ total score is composed of 22 items comprised of five subscales: Regimen Inconvenience (5 items), Lifestyle Flexibility (3 items), Glycemic Control (3 items), Hypoglycemic Control (5 items), and Insulin Delivery Device Satisfaction (6 items). Items use 7-point Likert scale responses, ranging from 1 (positive, e.g. "No bother at all") to 7 (negative, e.g. "A tremendous bother"), though the specific response labels vary by question. Items were reverse scored and transformed to range from 0 to 100. Higher scores indicate higher treatment satisfaction.
  score on a scale | 75.0 (14.4) | 75.6 (14.4) | 75.3 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: Time-in-serious Hypoglycemia
Description: % time spent less than 54 mg/dl averaged across all daily measures. For 6-month outcome, these data were averaged across two CGM sensors (placed at 6 and 6.5 months). For 12-month outcome, these data were from one CGM sensor placed at 11.5 months.
Time Frame: 6 and 12 months after randomization
Population: Randomized participants still on study with available CGM data at each time point
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 195 | 197
percentage of time
  6-month: number analyzed (Participants) | 194 | 196
  6-month | 3.6 (5.6) | 3.4 (4.3)
  12-month: number analyzed (Participants) | 172 | 184
  12-month | 2.4 (3.5) | 3.8 (5.5)
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 6-month (primary); Test type: Superiority; p = 0.43, Regression, Linear — Since this is one of two coprimary outcomes (this outcome and % time-in-range), a win (p<0.025 for benefit) on either outcome will be considered to be a positive trial; Multivariable generalized linear regression model adjusted for age at screening, study site, and % time in serious hypoglycemia at baseline
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 12-month; Test type: Superiority; p = 0.008, Regression, Linear — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Time-in-range (TIR)
Description: % time spent between 70 and 180mg/dl inclusive averaged across all daily measures. For 6-month outcome, these data were averaged across two CGM sensors (placed at 6 and 6.5 months). For 12-month outcome, these data were from one CGM sensor placed at 11.5 months.
Time Frame: 6 and 12 months after randomization
Population: Randomized participants still on study with available CGM data at each time point
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 195 | 197
percentage of time
  6-month: number analyzed (Participants) | 194 | 196
  6-month | 40.5 (18.4) | 38.1 (18.1)
  12-month: number analyzed (Participants) | 172 | 184
  12-month | 38.5 (20.1) | 37.7 (19.7)
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 6-month (primary); Test type: Superiority; p = 0.71, Regression, Linear — Since this is one of two coprimary outcomes (this outcome and % time in serious hypoglycemia), a win (p<0.025 for benefit) on either outcome will be considered to be a positive trial; Multivariable generalized linear regression model adjusted for age at screening, study site, and % TIR at baseline
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 12-month; Test type: Superiority; p = 0.64, Regression, Linear — [p-value comment as in outcome 2, analysis 1]; Multivariable generalized linear regression model adjusted for age at screening, study site, and % TIR at baseline

3. Secondary Outcome: Time-in-hypoglycemia
Description: % time spent less than 70mg/dl averaged across all daily measures. For 6-month outcome, these data were averaged across two CGM sensors (placed at 6 and 6.5 months). For 12-month outcome, these data were from one CGM sensor placed at 11.5 months.
Time Frame: 6 and 12 months after randomization
Population: Randomized participants still on study with available CGM data at each time point
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 195 | 197
percentage of time
  6-month: number analyzed (Participants) | 194 | 196
  6-month | 10.8 (9.5) | 10.2 (8.5)
  12-month: number analyzed (Participants) | 172 | 184
  12-month | 9.4 (10.4) | 11.2 (10.8)
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 6-month; Test type: Superiority; p = 0.54, Regression, Linear; Multivariable generalized linear regression model adjusted for age at screening, study site, and % time in hypoglycemia at baseline
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 12-month; Test type: Superiority; p = 0.07, Regression, Linear; [statistical method as in outcome 3, analysis 1]

4. Secondary Outcome: Time-above-range
Description: % time spent greater than 180mg/dl averaged across all daily measures. For 6-month outcome, these data were averaged across two CGM sensors (placed at 6 and 6.5 months). For 12-month outcome, these data were from one CGM sensor placed at 11.5 months.
Time Frame: 6 and 12 months after randomization
Population: Randomized participants still on study with available CGM data at each time point
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 195 | 197
percentage of time
  6-month: number analyzed (Participants) | 194 | 196
  6-month | 48.7 (22.7) | 51.8 (23.4)
  12-month: number analyzed (Participants) | 172 | 184
  12-month | 52.1 (24.9) | 51.1 (26.0)
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 6-month; Test type: Superiority; p = 0.58, Regression, Linear; Multivariable generalized linear regression model adjusted for age at screening, study site, and % time above range at baseline
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 12-month; Test type: Superiority; p = 0.21, Regression, Linear; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Nocturnal Hypoglycemic Events
Description: Number of events defined as ≥15 minutes in duration <70 mg/dL between midnight and 6:00 am; specifically, at least 2 sensor values <70 mg/dL that are ≥15 minutes apart plus no intervening values ≥70 mg/dL For 6-month outcome, these data were averaged across two CGM sensors (placed at 6 and 6.5 months). For 12-month outcome, these data were from one CGM sensor placed at 11.5 months.
Time Frame: 6 and 12 months after randomization
Population: Randomized participants still on study with available CGM data during nocturnal hours at each time point
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 195 | 196
number of events
  6-month: number analyzed (Participants) | 194 | 195
  6-month | 3.5 (2.6) | 3.6 (2.7)
  12-month: number analyzed (Participants) | 172 | 181
  12-month | 3.2 (2.7) | 4.2 (3.5)
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 6-month; Test type: Superiority; p = 0.70, Regression, Linear; Multivariable generalized linear regression model adjusted for age at screening, study site, and number of nocturnal events at baseline
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 12-month; Test type: Superiority; p = 0.02, Regression, Linear; [statistical method as in outcome 5, analysis 1]

6. Secondary Outcome: Glycemic Control (HbA1c)
Description: Mean HbA1c lab result reported as percent, which is typically how it is reported.
Time Frame: baseline, 3, 6, 9 and 12 months after randomization
Population: Randomized participants still on study with available HbA1c data at each time point
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 199 | 201
percent
  Baseline | 9.7 (2.8) | 9.9 (2.8)
  3-month: number analyzed (Participants) | 197 | 200
  3-month | 9.3 (2.5) | 9.4 (2.5)
  6-month: number analyzed (Participants) | 195 | 199
  6-month | 9.4 (2.3) | 9.5 (2.4)
  9-month: number analyzed (Participants) | 192 | 195
  9-month | 9.5 (2.1) | 9.4 (2.2)
  12-month: number analyzed (Participants) | 188 | 197
  12-month | 9.4 (2.3) | 9.4 (2.5)
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 6-month; Test type: Superiority; p = 0.81, Regression, Linear; Multivariable generalized linear regression model adjusted for age at screening, study site, and HbA1c at baseline
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 12-month; Test type: Superiority; p = 0.29, Regression, Linear; Multivariable generalized linear regression model adjusted for age at screening, study site, and HbA1c at baseline

7. Secondary Outcome: Rate of Severe Hypoglycemic Events
Description: Severe hypoglycemic events (requiring assistance of another person to correct) reported by participant per 1000 person-years
Time Frame: 6 and 12 months after randomization
Population: Randomized participants who knew whether or not they had an event at least one of the time points post-baseline/run-in phase.
Measure: Number (95% Confidence Interval); unit: events per 1000 person years
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 197 | 200
events per 1000 person years
  6-month | 0 [0 to 6.83] | 3.11 [0 to 8.54]
  12-month | 1.33 [0 to 4.20] | 1.41 [0 to 4.29]
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); Through 6-month; Test type: Superiority; p = 0.98, Negative Binomial Regression; Negative binomial regression model adjusted for age at screening and study site
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); Through 12-month; Test type: Superiority; p = 0.61, Negative Binomial Regression; Negative binomial regression model adjusted for age at screening and study site

8. Secondary Outcome: Rate of Diabetic Ketoacidosis (DKA)
Description: Hospitalization or Emergency Room Visit (serious adverse event) with primary diagnosis of Diabetic Ketoacidosis. This was measured by self-report and confirmed through review of hospital records
Time Frame: 6 and 12 months after randomization
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: events per 1000 person years
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 197 | 200
events per 1000 person years
  6-month | 0 [0 to 0] | 0 [0 to 0]
  12-month | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); Through 6-month; Test type: Superiority; p = 0.83, Negative Binomial Regression; Negative binomial regression model adjusted for age at screening and study site
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); Through 12-month; Test type: Superiority; p = 0.09, Negative Binomial Regression; Negative binomial regression model adjusted for age at screening and study site

9. Secondary Outcome: Pediatric Quality of Life Inventory 3.2 Diabetes Module (PedsQL 3.2 DM) Diabetes Symptoms Score
Description: Mean PedsQL 3.2 DM Diabetes Symptoms score. PedsQL 3.2 DM Diabetes Symptoms scale is composed of 15 items. All items use the same 5-point Likert response scale, with responses ranging from "never" (0) to "almost always" (4). Items are reverse scored and transformed on a scale ranging from 0 to 100. The score is the sum of all the items over the number of items answered. Higher scores indicate fewer diabetes symptoms and therefore improved diabetes-specific health-related quality of life (D-HRQoL).
Time Frame: Baseline and at 6 and 12 months after randomization
Population: Randomized participants still on study with available PedsQL data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline | 68.1 (14.7) | 69.3 (14.0)
  6-month: number analyzed (Participants) | 195 | 199
  6-month | 74.6 (14.4) | 75.2 (14.1)
  12-month: number analyzed (Participants) | 187 | 196
  12-month | 75.9 (15.1) | 76.9 (14.5)
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 6-month; Test type: Superiority; p = 0.95, Regression, Linear; Multivariable generalized linear regression model adjusted for age at screening, study site, and PedsQL 3.2 DM Diabetes Symptoms score at baseline
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 12-month; Test type: Superiority; p = 0.73, Regression, Linear; [statistical method as in outcome 9, analysis 1]

10. Secondary Outcome: Pediatric Quality of Life Inventory 3.2 Diabetes Module (PedsQL 3.2 DM) Diabetes Management Score
Description: Mean PedsQL 3.2 DM Diabetes Management score. PedsQL 3.2 DM Diabetes Management scale is composed of 18 items. All items use the same 5-point Likert response scale, with responses ranging from "never" (0) to "almost always" (4). Items are reverse scored and transformed on a scale ranging from 0 to 100. Higher scores indicate fewer diabetes management problems and therefore improved D-HRQoL.
Time Frame: Baseline and at 6 and 12 months after randomization
Population: Randomized participants still on study with available PedsQL data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline | 80.0 (14.3) | 81.5 (13.8)
  6-month: number analyzed (Participants) | 195 | 199
  6-month | 85.8 (11.7) | 85.7 (11.0)
  12-month: number analyzed (Participants) | 187 | 196
  12-month | 88.0 (11.0) | 88.8 (10.3)
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 6-month; Test type: Superiority; p = 0.81, Regression, Linear; Multivariable generalized linear regression model adjusted for age at screening, study site, and PedsQL 3.2 DM Diabetes Management score at baseline
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 12-month; Test type: Superiority; p = 0.44, Regression, Linear; [statistical method as in outcome 10, analysis 1]

11. Secondary Outcome: Insulin Treatment Satisfaction Questionnaire (ITSQ) Scores
Description: The ITSQ is composed of 22 items. A total 22-item score is reported, and the items are also divided into five subscales: Regimen Inconvenience (5 items), Lifestyle Flexibility (3 items), Glycemic Control (3 items), Hypoglycemic Control (5 items), and Insulin Delivery Device Satisfaction (6 items). Items use 7-point Likert scale responses, ranging from 1 (positive, e.g. "No bother at all") to 7 (negative, e.g. "A tremendous bother"), though the specific response labels vary by question. Items were reverse scored and transformed to range from 0 to 100. Higher scores indicate higher treatment satisfaction.
Time Frame: Baseline and at 6 and 12 months after randomization
Population: Randomized participants still on study with available ITSQ data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline | 75.0 (14.4) | 75.6 (14.4)
  6-month: number analyzed (Participants) | 195 | 199
  6-month | 84.1 (9.0) | 82.1 (11.1)
  12-month: number analyzed (Participants) | 187 | 196
  12-month | 87.1 (7.9) | 85.9 (8.6)
Statistical Analysis 1: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 6-month; Test type: Superiority; p = 0.04, Regression, Linear; Multivariable generalized linear regression model adjusted for age at screening, study site, and ITSQ at baseline
Statistical Analysis 2: Comparison: Glargine vs NPH or Premixed 70/30 (Human Insulin); 12-month; Test type: Superiority; p = 0.10, Regression, Linear; Multivariable generalized linear regression model adjusted for age at screening, study site, and ITSQ at baseline

ADVERSE EVENTS:
Time Frame: Adverse event were data collected through 12 months
Description: Adverse events were assessed periodically throughout a participant's time on study and entered into a standard questionnaire on an as-needed basis
Arm/Group | Glargine | NPH or Premixed 70/30 (Human Insulin)
All-Cause Mortality (participants affected / at risk) | 0/199 | 1/201
Serious Adverse Events (participants affected / at risk) | 5/199 | 13/201
Other Adverse Events (participants affected / at risk) | 33/199 | 33/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine (N=199) | NPH or Premixed 70/30 (Human Insulin) (N=201)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 1 (2) | 0 (0)
Encephalitis infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Other (Infections and infestations) | 0 (0) | 1 (1) — Severe Malaria
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glargine (N=199) | NPH or Premixed 70/30 (Human Insulin) (N=201)
Hypoglycemia (Metabolism and nutrition disorders) | 31 (31) | 21 (24)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Other (Endocrine disorders) | 2 (2) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-07-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT05614089/Prot_SAP_008.pdf
  • Informed Consent Form: Informed Consent_ Bangladesh site (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT05614089/ICF_005.pdf
  • Informed Consent Form: Informed Consent_ Tanzania site (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/89/NCT05614089/ICF_006.pdf